CLINICAL TRIAL: NCT05202652
Title: A Randomized, Placebo-controlled Prospective Trial for the Evaluation of Anti-oxidant, Anti-aging and Wellbeing Effects of a Novel Nutraceutical Formulation (HealthSpan)
Brief Title: Evaluation of Anti-oxidant, Anti-aging and Wellbeing Effects of a Novel Nutraceutical Formulation (HealthSpan)
Acronym: HealthSpan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hellenic Research Foundation (Other)
Collaborators: Theracell Advanced Biotechnology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HealthSpan Trial
Record Dates: First submitted 2021-12-22; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Aging; Well Aging; Oxidative Stress
Keywords: nutraceuticals; dietary supplements; antioxidant defense; proteostasis; well-being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The control group received a three month supply of 90 vegetal capsules of hydroxypropyl methylcellulose, each of them containing 455mg of the carrier substance (magnesium stearate)
  Interventions: Dietary Supplement: Placebo
- HealthSpan(HS) Group (Active Comparator): The HS group received a three month supply of 90 vegetal capsules of hydroxypropyl methylcellulose, each of them containing the 455mg of the mixture of the active compounds along with the carrier.
  Interventions: Dietary Supplement: HealthSpan

INTERVENTIONS:
Dietary Supplement: HealthSpan — The intervention was conducted on a group of healthy volunteers of age 29-85 with a once-daily administration of the oral capsule containing the active ingredients, for three consecutive months.
  Arms: HealthSpan(HS) Group
Dietary Supplement: Placebo — The intervention was conducted on a group of healthy volunteers of age 29-85 with a once-daily administration of the placebo, for three consecutive months.
  Arms: Control Group

SUMMARY:
The study was designed as a randomized, placebo-controlled trial with follow-up at 3 months. The study is in accordance with the Declaration of Helsinki and was approved by the Institutional Bioethical Committee of the National Hellenic Research Foundation. All the study participants received informative material, filled a questionnaire regarding the self-assessment of their health status and nutritional habits, and signed their written informed consent. In total, excluding the participants that did not return for the follow-up (dropouts), 122 apparently healthy volunteers of age 29-85 were followed, with 43 of them being randomly assigned in the placebo subgroup and 79 receiving the composition of the present invention.

DETAILED DESCRIPTION:
The study was designed as a randomized, placebo-controlled trial with follow-up at 3 months. The study is in accordance with the Declaration of Helsinki and was approved by the Institutional Bioethical Committee of the National Hellenic Research Foundation. All the study participants received informative material, filled a questionnaire regarding the self-assessment of their health status and nutritional habits, and signed their written informed consent. Patients eligible for the inclusion criteria were randomized into two groups: the group of healthy adult volunteers that received a capsule with the active formulation and those the received the placebo (a capsule with only the carrier substance magnesium stearate) In total, excluding the participants that did not return for the follow-up (dropouts), 122 apparently healthy volunteers of age 29-85 were followed, with 43 of them being randomly assigned in the placebo subgroup and 79 receiving the composition of the present invention.

ELIGIBILITY:
Inclusion Criteria:

* residence in the Athens metropolitan area
* age 29-85

Exclusion Criteria:

* diagnosed cancer, subjects that were under chemotherapy, therapy with biological factors and radiotherapy
* use of nutritional supplements during the clinical trial period
* diagnosed autoimmune diseases or other chronic diseases
* subjects that had lived less than 50% of their life in the country that is their current residence.

Ages: 29 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Effect of the formulation on oxidized proteins' levels | 3 months
  Oxidative stress states can be indicative of an impaired antioxidant defense. The study focused on the assessment of oxidative stress status by the protein carbonyls' levels before and after the intervention.

SECONDARY OUTCOMES:
Analysis of the effect of the formulation on oxidized proteins' levels adjusted for sex, age, and lifestyle habits of the sample as assessed in the study's questionnaire | 3 months
  Analysis adjusted for specific parameters to reveal potential confounders of the primary outcome of the intervention.
Correlation of levels of oxidized proteins and measured 20S proteasome levels | 3 months
  Oxidized proteins are the preferred substrates for enzymatic degradation by the proteasome. The study also investigated the interrelation between those two biomarkers in order to assess the effect of the intervention in proteasomal proteolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Eftathios Gonos, PhD, Principal Investigator — National Hellenic Research Foundation
Locations (1):
- Institute of Chemical Biology of National Hellenic Research Foundation, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Data of the study (statistical analysis, demographics) will be shared upon forthcoming publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after publication (spring 2022)
Access Criteria: PIs affiliated with Research Institutions and Universities

REFERENCES:
- [Background] Beckman KB, Ames BN. The free radical theory of aging matures. Physiol Rev. 1998 Apr;78(2):547-81. doi: 10.1152/physrev.1998.78.2.547. PMID 9562038
- [Background] Beekman M, Blanche H, Perola M, Hervonen A, Bezrukov V, Sikora E, Flachsbart F, Christiansen L, De Craen AJ, Kirkwood TB, Rea IM, Poulain M, Robine JM, Valensin S, Stazi MA, Passarino G, Deiana L, Gonos ES, Paternoster L, Sorensen TI, Tan Q, Helmer Q, van den Akker EB, Deelen J, Martella F, Cordell HJ, Ayers KL, Vaupel JW, Tornwall O, Johnson TE, Schreiber S, Lathrop M, Skytthe A, Westendorp RG, Christensen K, Gampe J, Nebel A, Houwing-Duistermaat JJ, Slagboom PE, Franceschi C; GEHA consortium. Genome-wide linkage analysis for human longevity: Genetics of Healthy Aging Study. Aging Cell. 2013 Apr;12(2):184-93. doi: 10.1111/acel.12039. Epub 2013 Feb 6. PMID 23286790
- [Background] Catalgol B, Ziaja I, Breusing N, Jung T, Hohn A, Alpertunga B, Schroeder P, Chondrogianni N, Gonos ES, Petropoulos I, Friguet B, Klotz LO, Krutmann J, Grune T. The proteasome is an integral part of solar ultraviolet a radiation-induced gene expression. J Biol Chem. 2009 Oct 30;284(44):30076-86. doi: 10.1074/jbc.M109.044503. Epub 2009 Aug 18. PMID 19690165
- [Background] Chondrogianni N, Tzavelas C, Pemberton AJ, Nezis IP, Rivett AJ, Gonos ES. Overexpression of proteasome beta5 assembled subunit increases the amount of proteasome and confers ameliorated response to oxidative stress and higher survival rates. J Biol Chem. 2005 Mar 25;280(12):11840-50. doi: 10.1074/jbc.M413007200. Epub 2005 Jan 20. PMID 15661736
- [Background] Gonos E. Proteasome activation as a novel anti-aging strategy. Free Radic Biol Med. 2014 Oct;75 Suppl 1:S7. doi: 10.1016/j.freeradbiomed.2014.10.842. Epub 2014 Dec 10. PMID 26461417
- [Background] Kapetanou M, Chondrogianni N, Petrakis S, Koliakos G, Gonos ES. Proteasome activation enhances stemness and lifespan of human mesenchymal stem cells. Free Radic Biol Med. 2017 Feb;103:226-235. doi: 10.1016/j.freeradbiomed.2016.12.035. Epub 2016 Dec 27. PMID 28034832
- [Background] Weber D, Stuetz W, Toussaint O, Debacq-Chainiaux F, Dolle MET, Jansen E, Gonos ES, Franceschi C, Sikora E, Hervonen A, Breusing N, Sindlinger T, Moreno-Villanueva M, Burkle A, Grune T. Associations between Specific Redox Biomarkers and Age in a Large European Cohort: The MARK-AGE Project. Oxid Med Cell Longev. 2017;2017:1401452. doi: 10.1155/2017/1401452. Epub 2017 Jul 19. PMID 28804532
- [Background] Santoro A, Pini E, Scurti M, Palmas G, Berendsen A, Brzozowska A, Pietruszka B, Szczecinska A, Cano N, Meunier N, de Groot CP, Feskens E, Fairweather-Tait S, Salvioli S, Capri M, Brigidi P, Franceschi C; NU-AGE Consortium. Combating inflammaging through a Mediterranean whole diet approach: the NU-AGE project's conceptual framework and design. Mech Ageing Dev. 2014 Mar-Apr;136-137:3-13. doi: 10.1016/j.mad.2013.12.001. Epub 2013 Dec 14. PMID 24342354
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. The hallmarks of aging. Cell. 2013 Jun 6;153(6):1194-217. doi: 10.1016/j.cell.2013.05.039. PMID 23746838
- [Background] Aunan JR, Watson MM, Hagland HR, Soreide K. Molecular and biological hallmarks of ageing. Br J Surg. 2016 Jan;103(2):e29-46. doi: 10.1002/bjs.10053. PMID 26771470
- [Background] Chondrogianni N, Voutetakis K, Kapetanou M, Delitsikou V, Papaevgeniou N, Sakellari M, Lefaki M, Filippopoulou K, Gonos ES. Proteasome activation: An innovative promising approach for delaying aging and retarding age-related diseases. Ageing Res Rev. 2015 Sep;23(Pt A):37-55. doi: 10.1016/j.arr.2014.12.003. Epub 2014 Dec 23. PMID 25540941
- [Background] Gonos ES, Kapetanou M, Sereikaite J, Bartosz G, Naparlo K, Grzesik M, Sadowska-Bartosz I. Origin and pathophysiology of protein carbonylation, nitration and chlorination in age-related brain diseases and aging. Aging (Albany NY). 2018 May 17;10(5):868-901. doi: 10.18632/aging.101450. PMID 29779015
- [Background] Athanasopoulou S, Chondrogianni N, Santoro A, Asimaki K, Delitsikou V, Voutetakis K, Fabbri C, Pietruszka B, Kaluza J, Franceschi C, Gonos ES. Beneficial Effects of Elderly Tailored Mediterranean Diet on the Proteasomal Proteolysis. Front Physiol. 2018 May 1;9:457. doi: 10.3389/fphys.2018.00457. eCollection 2018. PMID 29765333